CLINICAL TRIAL: NCT01835119
Title: Influence of Gum Chewing on Postoperative Bowel Activity After Complete Staging Surgery for Gynecological Malignancies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Medical Doctor, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gungorduk14
Record Dates: First submitted 2013-04-10; First posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Postoperative Ileus
Keywords: gynecological malignancies; postoperative; bowel activity; gum chewing
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chewing gum (Experimental): Gum type was standardized with all subjects receiving sugar-free peppermint-flavored gum.
  The patients in the chewing gum group, gum chewing began the morning of postoperative day 1. Patients chewed gum (one stick) 3 times daily in the morning, afternoon, and evening at least 5 min. The administration of the therapy was implemented by ward nursing staff and recorded in the patients file. All gum-chewing patients completed their course of gum chewing until bowel function.
  Interventions: Drug: gum
- control group (No Intervention): no gum

INTERVENTIONS:
Drug: gum — gum
  Arms: chewing gum

SUMMARY:
Postoperative ileus can cause the accumulation of secretions and gas, resulting in nausea, vomiting and abdominal distension and pain. Prolonged paralytic ileus is one of the commonest reasons for delayed recovery and discharge from hospital following abdominal surgery. Advances in surgical techniques and peri-operative management such as the use of laparoscopic surgery, thoracic epidural analgesia, early postoperative feeding and mobilization, amongst others, have been shown to help in the resolution of postoperative ileus.

Chewing gum, as a proxy for sham feeding, may accelerate the motility of the GI tract by stimulating the cephalic phase of digestion and eliciting the release of multiple promotility GI hormones. A number of small controlled studies evaluating the effect of chewing gum on postoperative intestinal recovery in patients undergoing colorectal surgery have been conducted. Decreased time for bowel function recovery and decreased hospital length of stay have not been consistently documented, possibly owing to the insufficient power of existing studies and study design issues. In addition, all previous studies have been limited by their use of sugarfree gum, containing known motility agents (eg, sorbitol).

In this study, gum chewing was studied for its effect on women with surgical staging for malignant gynecologic disease such as endometrial cancer, cervix cancer and ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women who would undergo surgical staging for malignant gynecologic disease such as endometrial cancer, cervix cancer and ovarian cancer were assessed for eligibility.

Exclusion Criteria:

* women who had thyroid diseases, inflammatory bowel disease, complaints of chronic constipation (defined as two or less bowel movements per week), had a history of prior abdominal bowel surgery, abdominal radiation, or neoadjuvant chemotherapy,
* need for intensive care more that 24 hours postoperatively, had nasogastric tube drainage beyond the first postoperative morning bowel anastomosis in relation to their operation during the surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
postoperative flatus pass time | an expected average of 48 hours
  The main outcome variable of the study was postoperative flatus pass time (hours from end of operation). Participants will be followed for the duration of the flatus pass time, an expected average of 48 hours

SECONDARY OUTCOMES:
duration of hospital stay | an expected average of 3 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
gastrointestinal disturbance | an expected average of 3 weeks
  gastrointestinal disturbance such as nausea, abdominal cramping, abdominal distension, rate of vomiting
time to first bowel movement | an expected average of 48 hours hours from end of operation
  time to first bowel movement (hours from end of operation).Participants will be followed for time to first bowel movement, an expected average of 48 hours hours from end of operation
Time to first defaecation | an expected average of 72 hours
  The main outcome variable of the study was postoperative flatus pass time (hours from end of operation).Participants will be followed for the duration of the first defaecation time, an expected average of 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Tepecik training and research hospital, Izmir, Tepecik, Turkey (Türkiye)